CLINICAL TRIAL: NCT07277439
Title: A Prospective, Open-label, Randomized, Controlled Phase II Clinical Trial Exploring the Efficacy and Safety of Thymosin Alpha 1 Combined With PD-1 Monoclonal Antibody and Neoadjuvant Chemoradiotherapy for cStage III Gastroesophageal Junction Adenocarcinoma
Brief Title: Phase II Trial of Neoadjuvant Thymalfasin, PD-1 Inhibitor, and Chemoradiotherapy for cStage III GEJ Adenocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Hao Xu, Professor, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-SR-275
Record Dates: First submitted 2025-07-02; First posted 2025-12-11 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Immunomodulation

STUDY DESIGN:
Intervention Model Description: Patients were randomly assigned preoperatively in a 1:2 ratio:
  Immunomodulation group (n=32): 3 cycles of slulimab combined with SOX combined with radiotherapy and 9 weeks of thymosin-based neoadjuvant therapy; Radiochemoimmunotherapy group (n=16): 3 cycles of slulimab combined with SOX combined with radiotherapy.
  Radiotherapy was initiated 2-5 days after the start of the second cycle of immunochemoimmunotherapy. A 5-10 mm extravasation was made from the endoscopically marked tumor boundary and adjacent metastatic lymph nodes to form a central tumor volume (CTV), and another 5-10 mm extravasation was made to form a partial tumor volume (PTV). The planned PTV treatment time was 44 Gy/22 fractions per minute (F), 5 fractions per week (F/W).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immunomodulation group (Experimental): Immunomodulation group (n=32): 3 cycles of slulimab combined with SOX combined with radiotherapy and 9 weeks of thymosin-based neoadjuvant therapy;
  Interventions: Other: Immunomodulation
- Radiochemoimmunotherapy group (Experimental): Radiochemoimmunotherapy group (n=16): 3 cycles of slulimab combined with SOX combined with radiotherapy.
  Interventions: Other: Radiochemoimmunotherapy

INTERVENTIONS:
Other: Radiochemoimmunotherapy — 3 cycles of slulimab combined with SOX combined with radiotherapy.
  Arms: Radiochemoimmunotherapy group
Other: Immunomodulation — 3 cycles of slulimab combined with SOX combined with radiotherapy and 9 weeks of thymosin-based neoadjuvant therapy;
  Arms: Immunomodulation group

SUMMARY:
This is a prospective, single-center, randomized controlled, phase II clinical trial. The study aims to enroll 48 patients with resectable, locally advanced gastroesophageal junction adenocarcinoma who have not received any treatment. After obtaining informed consent and meeting the inclusion/exclusion criteria, patients were randomly assigned preoperatively in a 1:2 ratio:

Immunomodulation group (n=32): 3 cycles of slulimab combined with SOX combined with radiotherapy and 9 weeks of neoadjuvant thymosin;

Radiochemoimmunotherapy group (n=16): 3 cycles of slulimab combined with SOX combined with radiotherapy;

Radiotherapy was initiated 2-5 days after the start of the second cycle of immunochemotherapy. A 5-10 mm extravasation was made from the endoscopically marked tumor boundary and adjacent metastatic lymph nodes to form a central tumor volume (CTV), and a 5-10 mm extravasation was made to form a partial tumor volume (PTV). The planned PTV treatment time was 44 Gy/22 fractions per minute (F), 5 fractions per week (F/W).

After neoadjuvant therapy, the efficacy of the therapy and the feasibility of radical D2 resection are assessed through imaging examinations. Efficacy evaluation is performed within 2 weeks of the completion of neoadjuvant therapy, and radical gastrectomy is performed within 4-6 weeks. Postoperative treatment is determined jointly by the clinician and the patient based on actual clinical practice.

The primary endpoint is the safety of neoadjuvant therapy: the incidence of ≥ grade 3 treatment-related adverse events (TRAEs) during the perioperative period (from the start of neoadjuvant therapy to one month postoperatively).

Safety assessment: Safety assessments are performed after each cycle of neoadjuvant therapy and 30 days postoperatively.

Event follow-up: Follow-up events are then conducted every 3 months for the first year postoperatively, and every 6 months for 1-2 years, up to 2 years postoperatively.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written informed consent provided.
2. Age ≥ 18 years and ≤ 80 years at enrollment.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0-2.
4. Life expectancy ≥ 6 months.
5. Diagnosis of gastric (G) or gastroesophageal junction (GEJ) adenocarcinoma by gastroscopy and histopathology. According to AJCC 8th edition staging, abdominal CT assessment confirms clinical stage cStage III (cT3-4aN1-3M0). For GEJ cancers, only Siewert type III and those Siewert type II cases not requiring combined thoracotomy are eligible.
6. Meets the diagnostic criteria for cachexia (based on Fearon's criteria): Either of the following criteria **combined with anorexia or evidence of systemic inflammation**:

   * Unintentional weight loss >5% within the past 6 months; OR
   * BMI <18.5 kg/m² and unintentional weight loss >2% within the past 6 months; OR
   * Appendicular skeletal muscle index meeting criteria for sarcopenia (male <7.26 kg/m²; female <5.45 kg/m²) and unintentional weight loss >2% within the past 6 months.
7. Prior to enrollment, a multidisciplinary assessment involving at least one gastrointestinal surgery attending physician and one radiologist confirms cStage III disease, eligibility for R0 resection with curative intent, patient's agreement to undergo radical surgery, and absence of surgical contraindications as judged by the surgeon.
8. No prior systemic anti-cancer therapy for the current disease, including surgery, radiotherapy, chemotherapy, immunotherapy, etc.
9. Adequate cardiac function to undergo curative-intent resection. Patients with underlying ischemic, valvular, or other significant heart disease should undergo preoperative evaluation by a cardiologist if clinically indicated.
10. Adequate organ function, meeting the following laboratory parameters (without supportive measures within specified timeframes):

    * Absolute neutrophil count (ANC) ≥1.5 × 10⁹/L (without granulocyte colony-stimulating factor support within 14 days).
    * Platelets ≥100 × 10⁹/L (without transfusion within 14 days).
    * Hemoglobin >8 g/dL (without transfusion or erythropoietin use within 14 days).
    * Total bilirubin ≤1.5 × upper limit of normal (ULN); OR total bilirubin >1.5 × ULN but direct bilirubin ≤ ULN.
    * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 × ULN.
    * Serum creatinine ≤1.5 × ULN AND calculated creatinine clearance (Cockcroft-Gault formula) ≥60 mL/min.
    * Adequate coagulation, defined as International Normalized Ratio (INR) or prothrombin time (PT) ≤1.5 × ULN.
    * Normal thyroid function, defined as thyroid-stimulating hormone (TSH) within normal range. If baseline TSH is outside normal range, subjects with total T3 (or FT3) and FT4 within normal range are eligible.
    * Myocardial enzymes within normal limits (subjects with isolated lab abnormalities judged by the investigator as clinically insignificant may be eligible).
11. For female patients:

    * Postmenopausal (defined as ≥1 year of amenorrhea without an alternative cause), OR surgically sterilized (removal of ovaries and/or uterus), OR, if of childbearing potential, must meet all the following:

      * Negative pregnancy test within 7 days prior to first dose.
      * Agreement to use highly effective contraception (annual failure rate <1%) or practice abstinence from heterosexual intercourse from signing informed consent until at least 120 days after last dose of investigational product and at least 9 months after surgery. Highly effective methods include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.
    * Must not be breastfeeding.
12. For male patients: Agreement to practice abstinence from heterosexual intercourse or use contraception with the following details: If partner is a woman of childbearing potential or is pregnant, the male patient must remain abstinent or use a condom from signing informed consent until at least 120 days after last dose of investigational product and at least 9 months after surgery. The reliability of sexual abstinence should be evaluated considering the study duration and the patient's preferences and lifestyle. Periodic abstinence (calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods.
13. The subject has read and fully understands the patient information, and has signed the informed consent form.

Exclusion Criteria

Subjects who meet any of the following criteria will be excluded from this study:

1. History of other malignancies within the past 5 years or concurrent malignancy. Exceptions include cured localized tumors such as basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, carcinoma in situ of the prostate, cervical carcinoma in situ, breast carcinoma in situ, Stage I lung cancer, Stage I colorectal cancer, etc.
2. Planned or prior organ or bone marrow transplantation.
3. Blood transfusion within 2 weeks prior to the first dose, history of bleeding, or any grade 3 or higher bleeding event (per CTCAE v5.0) within 4 weeks prior to screening.
4. Coagulation disorders or bleeding tendency (INR >1.5 times the upper limit of normal [ULN] without anticoagulant use). Patients receiving therapeutic anticoagulation with agents such as warfarin, heparin, or analogues. Prophylactic use of low-dose warfarin (1 mg orally, once daily) or low-dose aspirin (≤100 mg daily) is permitted if INR ≤1.5.
5. Arterial or venous thromboembolic events within 6 months prior to screening, such as cerebrovascular accident (including transient ischemic attack), deep vein thrombosis (except catheter-related thrombosis secondary to prior chemotherapy deemed resolved by the investigator), and pulmonary embolism.
6. Myocardial infarction within 6 months prior to the first dose, or poorly controlled arrhythmias (including QTc interval ≥450 ms for males or ≥470 ms for females, calculated using Fridericia's formula).
7. Cardiac insufficiency meeting NYHA Class III-IV criteria, or left ventricular ejection fraction (LVEF) <50% as measured by echocardiogram.
8. Urinalysis showing protein ≥++ and confirmed 24-hour urine protein quantification >1.0 g.
9. Clinically symptomatic pleural effusion or ascites requiring intervention.
10. Known human immunodeficiency virus (HIV) infection.
11. Active pulmonary tuberculosis.
12. Non-healing wounds or incompletely healed fractures.
13. History or current presence of interstitial lung disease, pneumoconiosis, radiation pneumonitis, drug-related pneumonia, severely impaired pulmonary function, or other conditions that may interfere with the detection or management of suspected drug-related pulmonary toxicity.
14. Known active or suspected autoimmune disease. Patients in a stable state of the disease at enrollment (not requiring systemic immunosuppressive therapy) are allowed.
15. History of severe chronic autoimmune diseases (e.g., systemic lupus erythematosus), inflammatory bowel disease (e.g., ulcerative colitis, Crohn's disease), chronic diarrheal diseases (e.g., irritable bowel syndrome), sarcoidosis, or tuberculosis. Patients with active hepatitis B, hepatitis C, or HIV infection are excluded. Non-severe, well-controlled immune disorders (e.g., dermatitis, arthritis, psoriasis) are allowed. Hepatitis B virus titer <500 copies/mL is allowed.
16. Requirement for systemic corticosteroid therapy (>10 mg/day prednisone equivalent) or other immunosuppressive medications within 14 days prior to the first dose or during the study. Topical, inhaled, or physiologic replacement steroid doses (≤10 mg/day prednisone equivalent) are permitted in the absence of active autoimmune disease.
17. Any active infection requiring systemic anti-infective therapy within 14 days prior to the first dose. Prophylactic antibiotic use (e.g., for urinary tract infection or COPD) is allowed.
18. Administration of live vaccines within 28 days prior to the first dose. Inactivated seasonal influenza vaccines are allowed.
19. Prior treatment with antibodies/drugs targeting immune checkpoints (e.g., PD-1, PD-L1, CTLA-4 inhibitors).
20. Concurrent participation in another interventional clinical trial. Participation in observational or surgical studies is allowed.
21. Known history of allergy or intolerance to any component of the investigational product(s).
22. History of alcohol abuse, drug abuse, or substance dependence. Patients who have ceased alcohol consumption are allowed.
23. Patients considered likely to be non-compliant with the study protocol, affecting efficacy or safety assessments, or those with incomplete data.
24. Pregnant or breastfeeding women.
25. Any condition affecting gastrointestinal absorption (e.g., dysphagia, prior gastrectomy, uncontrolled vomiting), ongoing tube feeding or parenteral nutrition, anorexia nervosa, anorexia due to psychiatric disorders, or inability to eat due to pain.
26. Current or planned use of other appetite-stimulating or weight-gaining medications (e.g., corticosteroids [except short-term dexamethasone during chemotherapy], androgens, progestins, thalidomide, olanzapine, anamorelin, or other appetite stimulants).
27. Cushing's syndrome, adrenal or pituitary insufficiency; poorly controlled diabetes mellitus.
28. Postmenopausal women with a history of abnormal vaginal bleeding within the past year; premenopausal women with a history of abnormal endometrial thickening (>15 mm) within the past year.
29. Any arterial thromboembolic event within 6 months prior to the first dose; Grade 3 or higher venous thromboembolic event per NCI CTCAE v5.0 requiring urgent intervention (e.g., pulmonary embolism, cardiac chamber embolism); transient ischemic attack, cerebrovascular accident, hypertensive crisis, or hypertensive encephalopathy; acute exacerbation of chronic obstructive pulmonary disease within 1 month prior to the first dose; uncontrolled hypertension (SBP ≥160 mmHg or DBP ≥100 mmHg despite oral antihypertensive medication).
30. History of severe bleeding tendency or coagulation dysfunction; clinically significant bleeding symptoms within 1 month prior to the first dose, including but not limited to gastrointestinal bleeding, hemoptysis (defined as coughing or spitting ≥1 teaspoon of fresh blood or small blood clots, or coughing blood without sputum; blood-tinged sputum is allowed), epistaxis (excluding minor nosebleeds and blood-tinged postnasal drip).
31. Any condition that may increase the risk associated with study participation or investigational product use, or other severe, acute, or chronic medical conditions that, in the investigator's judgment, make the patient unsuitable for the clinical study.
32. Any other circumstances deemed by the investigator to make the patient unsuitable for participation in this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-12-16 (Estimated); Primary Completion 2027-02-16 (Estimated); Study Completion 2029-02-16 (Estimated)

PRIMARY OUTCOMES:
Safety of neoadjuvant therapy | from the start of neoadjuvant therapy to one month postoperatively
  Perioperative period incidence of ≥ grade 3 treatment-related adverse events (TRAEs).

SECONDARY OUTCOMES:
Major Pathological Response (MPR) | from preoperative to 10 days postoperative
  For patients with surgically resectable gastric cancer after neoadjuvant therapy, the proportion of patients with less than 10% residual tumor cells in the primary site.
Tumor Regression Grade (TRG) | from preoperative to 10 days postoperative
  It is intended to grade the pathological response of tumor after neoadjuvant therapy and generally divide the grade mainly according to the proportion of fibrosis and residual tumor in the tumor. In this study, Becker criteria are used to grade TGR as follows: TRG1a (no residual tumor), equivalent to pCR; TRG1b (< 10% residual tumor); TRG2 (10% to 50% residual tumor); and TRG3 (> 50% residual tumor).
Objective Response Rate (ORR) | before surgery
  It refers to the proportion of patients whose tumor shrinks to a certain extent and remains for a certain period of time, including CR (Complete Response) and PR (Partial Response) cases. Objective tumor response will be assessed using Response Evaluation Criteria in Solid Tumors (RECIST 1.1 criteria).
Disease-free Survival (DFS) | 2 years after surgery
  Disease-free survival refers to the time from the start of randomization to disease recurrence or death due to disease progression. DFS will be defined as the last date the patient is last confirmed to be disease-free survival if the patient does not experience disease progression during the study.
R0 resection rate | from preoperative to 10 days postoperative
  R0 resection rate refers to the proportion of patients who complete R0 resection in surgically resectable patients after neoadjuvant therapy.
treatment-related adverse event (TRAE) | from the start of neoadjuvant therapy to 30 days after surgery
  incidence of treatment-related adverse event
Complete pathological response (pCR) rate | from surgery to 1 month after surgery
  Defined as the proportion of subjects who have no residual surviving tumor cells under microscopic examination and are negative for lymph nodes;

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Nanjing Medical Unviersity, Nanjing, Jiangsu, China